CLINICAL TRIAL: NCT03591445
Title: Is Bronchoscopy Necessary in the Preoperative Workup of Ground Glass Opacity Featured Lung Cancer?
Brief Title: Is Bronchoscopy Necessary in the Preoperative Workup of GGO Lung Cancer?(ECTOP-1005)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Henan Cancer Hospital (Other Government); Anhui Chest Hospital (Other); Shanghai Zhongshan Hospital (Other); Affiliated Hospital of Jiangnan University (Other); Jilin Provincial Tumor Hospital (Other); Guanxian Central Hospital of Shandong Province (Unknown); The Third people's Hospital of Jieyang (Unknown); Queen Mary Hospital, Hong Kong (Other); Jiangdu people's hospital of Yangzhou Jiangsu Province (Unknown)
Responsible Party: Principal Investigator, Haiquan Chen, Director of Department of thoracic surgery and multidisciplinary group of thoracic oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Fudan_bronchoscopy
Record Dates: First submitted 2018-07-07; First posted 2018-07-19 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Pulmonary Nodule, Solitary
MeSH Terms: conditions — Solitary Pulmonary Nodule

STUDY DESIGN:
Intervention Model Description: We hypothesized incidence rate that bronchoscopic findings would have changed the rate of established surgical plans as less than 2.0% (P0), then preoperative bronchoscopy examination would have limited impact on the surgical plan for GGO featured lung cancer; If bronchoscopic findings would have changed the rate of established surgical plans as more than 4.0% (P1), then bronchoscopy examination would be regarded as one routine preoperative work-up. Null hypothesis: H0: P≤P0; Alternative hypothesis: HA: P ≥ P1. α = 0.05, 1-β = 0.9. Using Simon's two-stage approach, the first phase enrolled 612 patients. If ≥18 patients supported the alternative hypothesis, they entered the second phase, otherwise the trial was terminated; the second phase enrolled 451 patients. If the patient number who eventually changes the surgical plan is ≤27, the null hypothesis is accepted, that preoperative bronchoscopy examination would be unnecessary for GGO featured lung cancer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental：Bronchoscopy (Experimental): Patients with ground glass opacity featured lung cancer who are candidates for surgeyr received the bronchoscopy examination before surgery.
  Interventions: Device: Flexible Bronchoscopy

INTERVENTIONS:
Device: Flexible Bronchoscopy — Flexible Bronchoscopy

SUMMARY:
This study is one of Eastern Cooperative Thoracic Oncology Projects (ECTOP-1005). It aims to evaluate the role of flexible bronchoscopy in the pre-operative workup of ground glass opacity featured lung cancer. All enrolled patients receive the flexible bronchoscopy examination before surgery. Investigators observe the intra-bronchial findings of bronchoscopy and the impact of these findings on established surgical plan.

DETAILED DESCRIPTION:
The appropriateness of routine use of bronchoscopy in the operative workup of a solitary pulmonary nodule（SPN） is debatable. Options expressed in the literature vary from routine preoperative bronchoscopy having no role in obtaining tissue diagnosis in small SPNs to it begin very useful in determining underlying etiology and surgical strategy. The American College of Chest Physicians（ACCP）guidelines recommend bronchoscopy only if air-bronchogram is present or if operator has expertise with newer guided techniques. Previous study showed that bronchoscopy is not indicated in SPNs that present with ground-glass opacity on CT. The purpose of this analysis is to define that role by examining in GGO patients （1）intra-bronchial findings （2）impact of these findings on established surgical plan.

ELIGIBILITY:
Inclusion Criteria:

* Ground glass opacity pulmonary nodule diagnosed by thoracic CT
* karnofsky performance status ≥60
* No surgical contraindication
* Patients who sign the informed consent
* Pre-operation clinical stage :T1abcN0M0
* Age:18-80 years old

Exclusion Criteria:

* Central lung tumor diagnosed by CT
* Tracheal or bronchus deformity diagnosed by CT
* Tracheal or bronchus disease history
* Severe smoking history （smoking index ≥400/year）

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 615 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence rate that established surgical plan is changed by positive intra-bronchial findings | about 14 days
  The number of patients （surgical plan is changed by positive intra-bronchial findings） /Total number of patients

SECONDARY OUTCOMES:
rate of positive intra-bronchial findings | about 14 days
  the number of patients with positive intra-bronchial findings / total number of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China